CLINICAL TRIAL: NCT00782210
Title: Randomised, Double-blind, Placebo-controlled, Parallel Group Study to Assess the Efficacy and Safety of 48 Weeks of Once Daily Treatment of Orally Inhaled BI 1744 CL (5 mcg [2 Actuations of 2.5 mcg] and 10 mcg [2 Actuations of 5 mcg]) Delivered by the Respimat® Inhaler, in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: 12 / 48 Week Pivotal PFT vs PBO in COPD I
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1222.11; 2008-003647-36 (EudraCT Number: EudraCT)
Record Dates: First submitted 2008-10-29; First posted 2008-10-31 (Estimated); Results first posted 2014-04-30 (Estimated); Last update posted 2014-06-09 (Estimated); Status verified 2014-03

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — olodaterol

ARMS (3):
- Olodaterol (BI 1744) Low (Experimental): Low dose inhaled orally once daily from the Respimat inhaler
  Interventions: Drug: Olodaterol (BI1744)
- Olodaterol (BI 1744) High (Experimental): High dose inhaled orally once daily from the Respimat inhaler
  Interventions: Drug: Olodaterol (BI1744)
- Placebo (Placebo Comparator): Olodaterol (BI1744) placebo inhaled orally once daily from the Respimat inhaler
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Olodaterol (BI1744) — Comparison of low and high doses on efficacy and safety in COPD patients
  Arms: Olodaterol (BI 1744) Low
Drug: Olodaterol (BI1744) — Comparison of low and high doses on efficacy and safety in COPD patients
  Arms: Olodaterol (BI 1744) High
Drug: placebo — Olodaterol (BI1744) placebo inhaled orally once daily from the Respimat inhaler
  Arms: Placebo

SUMMARY:
This primary objective of this study is to compare two doses of BI 1744 CL inhalation solution delivered by the Respimat® inhaler once daily to placebo in patients with chronic obstructive pulmonary disease (COPD).

The safety of BI 1744 CL inhalation solution delivered through the Respimat inhaler will also be compared to placebo.

ELIGIBILITY:
Inclusion criteria:

* All patients must have a diagnosis of chronic obstructive pulmonary disease
* Male or female patients, 40 years of age or older Patients must be current or ex-smokers with a smoking history of more than 10 pack years Post bronchodilator FEV1 <80% predicted and post-bronchodilator FEV1/FVC <70%

Exclusion criteria:

* Patients with a significant disease other than COPD
* Patients with a history of asthma
* Patients with any of the following conditions:

a history of myocardial infarction within 1 year of screening visit (Visit 1) unstable or life-threatening cardiac arrhythmia. have been hospitalized for heart failure within the past year. known active tuberculosis a malignancy for which patient has undergone resection, radiation therapy or chemotherapy within last five years (patients with treated basal cell carcinoma are allowed) a history of life-threatening pulmonary obstruction a history of cystic fibrosis

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 625 (Actual)
Dates: Start 2008-11; Primary Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (54):
- United States (21):
  - 1222.11.1122 Boehringer Ingelheim Investigational Site, Jasper, Alabama
  - 1222.11.1116 Boehringer Ingelheim Investigational Site, Berkeley, California
  - 1222.11.1121 Boehringer Ingelheim Investigational Site, Los Angeles, California
  - 1222.11.1111 Boehringer Ingelheim Investigational Site, Fort Collins, Colorado
  - 1222.11.1117 Boehringer Ingelheim Investigational Site, Stamford, Connecticut
  - 1222.11.1110 Boehringer Ingelheim Investigational Site, DeLand, Florida
  - 1222.11.1106 Boehringer Ingelheim Investigational Site, Coeur d'Alene, Idaho
  - 1222.11.1108 Boehringer Ingelheim Investigational Site, Evansville, Indiana
  - 1222.11.1109 Boehringer Ingelheim Investigational Site, Bowling Green, Kentucky
  - 1222.11.1113 Boehringer Ingelheim Investigational Site, St Louis, Missouri
  - 1222.11.1115 Boehringer Ingelheim Investigational Site, Larchmont, New York
  - 1222.11.1120 Boehringer Ingelheim Investigational Site, Toledo, Ohio
  - 1222.11.1105 Boehringer Ingelheim Investigational Site, Oklahoma City, Oklahoma
  - 1222.11.1112 Boehringer Ingelheim Investigational Site, Charleston, South Carolina
  - 1222.11.1119 Boehringer Ingelheim Investigational Site, Greer, South Carolina
  - 1222.11.1102 Boehringer Ingelheim Investigational Site, Union, South Carolina
  - 1222.11.1124 Boehringer Ingelheim Investigational Site, Killeen, Texas
  - 1222.11.1101 Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - 1222.11.1103 Boehringer Ingelheim Investigational Site, Spokane, Washington
  - 1222.11.1114 Boehringer Ingelheim Investigational Site, Spokane, Washington
  - 1222.11.1123 Boehringer Ingelheim Investigational Site, Tacoma, Washington
- Australia (5):
  - 1222.11.1143 Boehringer Ingelheim Investigational Site, Concord, New South Wales
  - 1222.11.1145 Boehringer Ingelheim Investigational Site, Glebe, New South Wales
  - 1222.11.1144 Boehringer Ingelheim Investigational Site, Westmead, New South Wales
  - 1222.11.1142 Boehringer Ingelheim Investigational Site, Toorak Gardens, South Australia
  - 1222.11.1141 Boehringer Ingelheim Investigational Site, Woodville, South Australia
- China (11):
  - 1222.11.1166 Boehringer Ingelheim Investigational Site, Beijing
  - 1222.11.1171 Boehringer Ingelheim Investigational Site, Changsha
  - 1222.11.1170 Boehringer Ingelheim Investigational Site, Chengdu
  - 1222.11.1169 Boehringer Ingelheim Investigational Site, Chongqing
  - 1222.11.1172 Boehringer Ingelheim Investigational Site, Dalian
  - 1222.11.1163 Boehringer Ingelheim Investigational Site, Guangzhou
  - 1222.11.1167 Boehringer Ingelheim Investigational Site, Nanjing
  - 1222.11.1164 Boehringer Ingelheim Investigational Site, Shanghai
  - 1222.11.1165 Boehringer Ingelheim Investigational Site, Shanghai
  - 1222.11.1173 Boehringer Ingelheim Investigational Site, Shenyang
  - 1222.11.1168 Boehringer Ingelheim Investigational Site, Xi'an
- Germany (8):
  - 1222.11.1151 Boehringer Ingelheim Investigational Site, Berlin
  - 1222.11.1156 Boehringer Ingelheim Investigational Site, Berlin
  - 1222.11.1157 Boehringer Ingelheim Investigational Site, Erfurt
  - 1222.11.1154 Boehringer Ingelheim Investigational Site, Halle
  - 1222.11.1153 Boehringer Ingelheim Investigational Site, Kassel
  - 1222.11.1158 Boehringer Ingelheim Investigational Site, Oschersleben
  - 1222.11.1152 Boehringer Ingelheim Investigational Site, Potsdam
  - 1222.11.1155 Boehringer Ingelheim Investigational Site, Weinheim
- New Zealand (4):
  - 1222.11.1138 Boehringer Ingelheim Investigational Site, Hamilton
  - 1222.11.1139 Boehringer Ingelheim Investigational Site, Otahuhu
  - 1222.11.1136 Boehringer Ingelheim Investigational Site, Tauranga
  - 1222.11.1137 Boehringer Ingelheim Investigational Site, Wellington
- Taiwan (5):
  - 1222.11.1180 Boehringer Ingelheim Investigational Site, Changhua
  - 1222.11.1181 Boehringer Ingelheim Investigational Site, Chiayi City
  - 1222.11.1179 Boehringer Ingelheim Investigational Site, Taichung
  - 1222.11.1177 Boehringer Ingelheim Investigational Site, Taipei
  - 1222.11.1178 Boehringer Ingelheim Investigational Site, Taipei

REFERENCES:
- [Derived] Singh D, Wedzicha JA, Siddiqui S, de la Hoz A, Xue W, Magnussen H, Miravitlles M, Chalmers JD, Calverley PMA. Blood eosinophils as a biomarker of future COPD exacerbation risk: pooled data from 11 clinical trials. Respir Res. 2020 Sep 17;21(1):240. doi: 10.1186/s12931-020-01482-1. PMID 32943047
- [Derived] Andreas S, Bothner U, de la Hoz A, Kloer I, Trampisch M, Alter P. A Post Hoc Holter ECG Analysis of Olodaterol and Formoterol in Moderate-to-Very-Severe COPD. Int J Chron Obstruct Pulmon Dis. 2020 Aug 10;15:1955-1965. doi: 10.2147/COPD.S246353. eCollection 2020. PMID 32848381
- [Derived] Andreas S, Bothner U, Trampisch M, Haensel M, Buhl R, Alter P. Effect of long-acting beta2-agonists olodaterol and formoterol on heart rate and blood pressure in chronic obstructive pulmonary disease patients. Pulm Pharmacol Ther. 2018 Oct;52:1-6. doi: 10.1016/j.pupt.2018.08.002. Epub 2018 Aug 2. PMID 30077810
- [Derived] Ferguson GT, Feldman GJ, Hofbauer P, Hamilton A, Allen L, Korducki L, Sachs P. Efficacy and safety of olodaterol once daily delivered via Respimat(R) in patients with GOLD 2-4 COPD: results from two replicate 48-week studies. Int J Chron Obstruct Pulmon Dis. 2014 Jun 16;9:629-45. doi: 10.2147/COPD.S61717. eCollection 2014. PMID 24966672

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Matching Placebo delivered by the Respimat Inhaler.
- Olodaterol (Olo) 5 mcg qd: Olodaterol 5 mcg qd (morning) delivered by the Respimat Inhaler.
- Olodaterol (Olo) 10 mcg qd: Olodaterol 10 mcg qd (morning) delivered by the Respimat Inhaler.
Period: Overall Study
Arm/Group | Placebo | Olodaterol (Olo) 5 mcg qd | Olodaterol (Olo) 10 mcg qd
Started | 209 | 208 | 207
Completed | 159 | 173 | 172
Not Completed | 50 | 35 | 35
Not completed — Adverse Event | 21 | 17 | 16
Not completed — Lost to Follow-up | 2 | 1 | 2
Not completed — Withdrawal by Subject | 11 | 8 | 11
Not completed — Non compliance with protocol | 0 | 3 | 2
Not completed — Lack of Efficacy | 13 | 4 | 1
Not completed — Other reason not described above | 3 | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Olo 5 mcg qd: Olodaterol 5 mcg qd (morning) delivered by the Respimat Inhaler.
- Olo 10 mcg qd: Olodaterol 10 mcg qd (morning) delivered by the Respimat Inhaler.
- Total: Total of all reporting groups
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Total
Number analyzed (Participants) | 209 | 208 | 207 | 624
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.8 (8.5) | 64.0 (8.6) | 65.0 (8.2) | 64.9 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 58 | 52 | 167
  Male | 152 | 150 | 155 | 457
Tiotropium (Tio) Use Stratum [Number; unit: Number of participants]
  Non-tiotropium | 160 | 161 | 156 | 477
  Tiotropium | 49 | 47 | 51 | 147

OUTCOME MEASURES:

1. Primary Outcome: Forced Expiratory Volume in One Second (FEV1) Area Under Curve 0-3 Hour (h) (AUC 0-3h) Response at Day 85 (12 Weeks)
Description: Response was defined as change from baseline. Baseline FEV1 was defined as the mean of the -1 h and -10 min measurements performed just prior to administration of the first am dose of randomized treatment. Means are adjusted using a mixed effects model with treatment (trt), tio stratum, visit, trt-by-visit interaction as fixed categorical effects, baseline and baseline-by-visit interaction as fixed continuous covariates and patient as random effect. FEV1 AUC 0-3h was calculated from 0-3 hours post-dose using the trapezoidal rule, divided by the observation time (3h) to report in litres.
Time Frame: 1 hour (h) and 10 minutes (min) prior to dose on the first day of randomized treatment (baseline) to -10 min, 5 min, 15 min, 30 min, 1 h, 2 h, and 3 h relative to dose on Day 85
Population: Full analysis set (FAS). FAS is defined as all randomized patients who received at least one dose of treatment and had both baseline data and at least one post-baseline measurement at or before Day 85 (12 weeks) for either co-primary efficacy variable.
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 208 | 206 | 206
Liter | -0.007 (0.014) | 0.165 (0.014) | 0.169 (0.014)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effects model with trt,tio stratum,visit,trt-by-visit as fixed effects,baseline, baseline-by-visit as fixed covariates, patient as random effect; Mean Difference (Final Values) = 0.172, 95% CI [0.135 to 0.209], Standard Error of Mean 0.019 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.176, 95% CI [0.139 to 0.214], Standard Error of Mean 0.019 — Olo 10 mcg qd minus Placebo

2. Primary Outcome: Trough FEV1 Response at Day 85 (12 Weeks)
Description: Response was defined as change from baseline. Baseline trough FEV1 was defined as the mean of the -1 hour and -10 minute measurements performed just prior to first dose of randomized treatment. Trough FEV1 is defined as the FEV1 performed at -10 mins prior to study drug inhalation as the end of the dosing interval or the mean of -1h and -10 min FEV1s if both available. Means are adjusted using a mixed effects model with treatment (trt), tio stratum, visit, trt-by-visit as fixed categorical effects, baseline and baseline-by-visit as fixed continuous covariates and patient as random effect.
Time Frame: 1 h and 10 min prior to dose on the first day of randomized treatment (baseline) and -1 h and - 10 mins prior to study drug at Day 85.
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 200 | 199 | 202
Liter | -0.041 (0.014) | 0.050 (0.014) | 0.060 (0.014)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.091, 95% CI [0.054 to 0.128], Standard Error of Mean 0.019 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.101, 95% CI [0.064 to 0.137], Standard Error of Mean 0.019 — Olo 10 mcg qd minus Placebo

3. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) Area Under Curve 0-12 h (AUC 0-12h) Response at Day 85 (12 Weeks)
Description: Response was defined as change from baseline. Study baseline FEV1 was defined as the mean of the available pre-dose FEV1 values prior to the first dose of randomized treatment. Means are adjusted using a non-mixed effects model with treatment (trt), tio stratum, baseline as fixed effects. FEV1 AUC 0-12h was calculated from 0-12 hours post-dose using the trapezoidal rule, divided by the observation time (12h) to report in litres.
Time Frame: 1 hour (h) and 10 minutes (min) prior to dose on first day of randomized treatment (baseline) and -1h and -10 min, 5 min, 15 min, 30 min, 1h, 2h, 3h, 4h, 5h, 6h, 8h, 10h, 12h relative to dose at Day 85 (12 weeks)
Population: Patients in FAS with spirometry data after 3 hours at Visit 5 (12-hour pulmonary function test set)
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 71 | 85 | 85
Liter | -0.029 (0.025) | 0.144 (0.022) | 0.139 (0.022)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, ANCOVA; Treatment, tiotropium stratum and baseline as fixed effects; Mean Difference (Final Values) = 0.173, 95% CI [0.113 to 0.233], Standard Error of Mean 0.031 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Treatment, tiotropium stratum and baseline as fixed effects; Mean Difference (Final Values) = 0.169, 95% CI [0.108 to 0.229], Standard Error of Mean 0.031 — Olo 10 mcg qd minus Placebo

4. Secondary Outcome: Forced Expiratory Volume in One Second (FEV1) Area Under Curve 0-3 Hour (h) (AUC 0-3h) Response at Day 1
Description: Response was defined as change from baseline. Baseline FEV1 was defined as the mean of the -1 h and -10 min measurements performed just prior to administration of the first dose of randomized treatment. Means are adjusted using a mixed effects model with treatment (trt), tio stratum, visit, trt-by-visit interaction as fixed categorical effects, baseline and baseline-by-visit interaction as fixed continuous covariates and patient as random effect. FEV1 AUC 0-3h was calculated from 0-3 hours post-dose using the trapezoidal rule, divided by the observation time (3h) to report in litres.
Time Frame: 1 hour (h) and 10 minutes (min) prior to dose on the first day of randomized treatment (baseline) to -10 min, 5 min, 15 min, 30 min, 1 h, 2 h, and 3 h relative to dose at day 1
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Groups:
- Olo 10 mcg qd: Olodaterol 10 mcg qd (morning delivered by the Respimat Inhaler.
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 208 | 206 | 206
Liter | 0.024 (0.014) | 0.189 (0.014) | 0.199 (0.014)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.165, 95% CI [0.128 to 0.201], Standard Error of Mean 0.019 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.175, 95% CI [0.139 to 0.212], Standard Error of Mean 0.019 — Olo 10 mcg qd minus Placebo

5. Secondary Outcome: Forced Expiratory Volume in One Second (FEV1) Area Under Curve 0-3 Hour (h) (AUC 0-3h) Response After 2 Weeks
Description: as for outcome 4
Time Frame: 1 hour (h) and 10 minutes (min) prior to dose on the first day of randomized treatment (baseline) to -10 min, 5 min, 15 min, 30 min, 1 h, 2 h, and 3 h relative to dose after 2 weeks
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 208 | 206 | 206
Liter | -0.000 (0.014) | 0.180 (0.014) | 0.192 (0.014)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.181, 95% CI [0.144 to 0.217], Standard Error of Mean 0.019 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.192, 95% CI [0.156 to 0.229], Standard Error of Mean 0.019 — Olo 10 mcg qd minus Placebo

6. Secondary Outcome: Forced Expiratory Volume in One Second (FEV1) Area Under Curve 0-3 Hour (h) (AUC 0-3h) Response After 6 Weeks
Description: as for outcome 4
Time Frame: 1 hour (h) and 10 minutes (min) prior to dose on the first day of randomized treatment (baseline) to -1h, -10 min, 5 min, 15 min, 30 min, 1 h, 2 h, and 3 h relative to dose after 6 weeks
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 208 | 206 | 206
Liter | -0.001 (0.014) | 0.169 (0.014) | 0.165 (0.014)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.170, 95% CI [0.133 to 0.207], Standard Error of Mean 0.019 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.167, 95% CI [0.130 to 0.204], Standard Error of Mean 0.019 — Olo 10 mcg qd minus Placebo

7. Secondary Outcome: Forced Expiratory Volume in One Second (FEV1) Area Under Curve 0-3 Hour (h) (AUC 0-3h) Response After 24 Weeks
Description: as for outcome 4
Time Frame: 1 hour (h) and 10 minutes (min) prior to dose on the first day of randomized treatment (baseline) to -10 min, 5 min, 15 min, 30 min, 1 h, 2 h, and 3 h relative to dose after 24 weeks
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 208 | 206 | 206
Liter | -0.18 (0.014) | 0.156 (0.014) | 0.143 (0.014)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.174, 95% CI [0.136 to 0.212], Standard Error of Mean 0.019 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.161, 95% CI [0.123 to 0.199], Standard Error of Mean 0.019 — Olo 10 mcg qd minus Placebo

8. Secondary Outcome: Forced Expiratory Volume in One Second (FEV1) Area Under Curve 0-3 Hour (h) (AUC 0-3h) Response After 48 Weeks
Description: as for outcome 4
Time Frame: 1 hour (h) and 10 minutes (min) prior to dose on the first day of randomized treatment (baseline) to -10 min, 5 min, 15 min, 30 min, 1 h, 2 h, and 3 h relative to dose after 48 weeks
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 208 | 206 | 206
Liter | -0.043 (0.014) | 0.130 (0.014) | 0.126 (0.014)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.173, 95% CI [0.134 to 0.211], Standard Error of Mean 0.019 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.169, 95% CI [0.131 to 0.208], Standard Error of Mean 0.020 — Olo 10 mcg qd minus Placebo

9. Secondary Outcome: Trough FEV1 Response After 2 Weeks
Description: Response was defined as change from baseline. Baseline trough FEV1 was defined as the mean of the -1 hour and -10 minute measurements performed just prior to first dose of randomized treatment. Trough FEV1 is defined as the FEV1 performed a -10 mins prior to study drug inhalation as the end of the dosing interval or the mean of -1h and -10 min FEV1s if both available. Means are adjusted using a mixed effects model with treatment (trt), tio stratum, visit, trt-by-visit as fixed categorical effects, baseline and baseline-by-visit as fixed continuous covariates and patient as random effect.
Time Frame: 1 h and 10 min prior to dose on the first day of randomized treatment (baseline) and -1 h (if available) and - 10 mins prior to study drug after 2 weeks
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 200 | 199 | 202
Liter | -0.019 (0.014) | 0.076 (0.014) | 0.091 (0.014)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.095, 95% CI [0.059 to 0.131], Standard Error of Mean 0.018 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.111, 95% CI [0.075 to 0.147], Standard Error of Mean 0.018 — Olo 10 mcg qd minus Placebo

10. Secondary Outcome: Trough FEV1 Response After 6 Weeks
Description: as for outcome 2
Time Frame: 1 h and 10 min prior to dose on the first day of randomized treatment (baseline) and -1 h (if available) and - 10 mins prior to study drug after 6 weeks
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 200 | 199 | 202
Liter | -0.022 (0.014) | 0.073 (0.014) | 0.069 (0.014)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.095, 95% CI [0.059 to 0.131], Standard Error of Mean 0.019 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.091, 95% CI [0.054 to 0.127], Standard Error of Mean 0.019 — Olo 10 mcg qd minus Placebo

11. Secondary Outcome: Trough FEV1 Response After 18 Weeks
Description: as for outcome 2
Time Frame: 1 h and 10 min prior to dose on the first day of randomized treatment (baseline) and -1 h (if available) and - 10 mins prior to study drug after 18 weeks
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 200 | 199 | 202
Liter | -0.042 (0.014) | 0.056 (0.014) | 0.059 (0.014)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.098, 95% CI [0.061 to 0.135], Standard Error of Mean 0.019 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.101, 95% CI [0.064 to 0.138], Standard Error of Mean 0.019 — Olo 10 mcg qd minus Placebo

12. Secondary Outcome: Trough FEV1 Response After 24 Weeks
Description: as for outcome 2
Time Frame: 1 h and 10 min prior to dose on the first day of randomized treatment (baseline) and -1 h (if available) and - 10 mins prior to study drug after 24 weeks
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 200 | 199 | 202
Liter | -0.050 (0.014) | 0.036 (0.014) | 0.039 (0.014)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.086, 95% CI [0.049 to 0.123], Standard Error of Mean 0.019 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.089, 95% CI [0.051 to 0.126], Standard Error of Mean 0.019 — Olo 10 mcg qd minus Placebo

13. Secondary Outcome: Trough FEV1 Response After 32 Weeks
Description: as for outcome 2
Time Frame: 1 h and 10 min prior to dose on the first day of randomized treatment (baseline) and -1 h (if available) and - 10 mins prior to study drug after 32 weeks
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 200 | 199 | 202
Liter | -0.051 (0.014) | 0.041 (0.014) | 0.034 (0.014)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.092, 95% CI [0.054 to 0.130], Standard Error of Mean 0.019 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.085, 95% CI [0.048 to 0.123], Standard Error of Mean 0.019 — Olo 10 mcg qd minus Placebo

14. Secondary Outcome: Trough FEV1 Response After 40 Weeks
Description: as for outcome 2
Time Frame: 1 h and 10 min prior to dose on the first day of randomized treatment (baseline) and -1 h (if available) and - 10 mins prior to study drug after 40 weeks
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 200 | 199 | 202
Liter | -0.061 (0.014) | 0.046 (0.014) | 0.044 (0.014)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.107, 95% CI [0.069 to 0.145], Standard Error of Mean 0.019 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.105, 95% CI [0.068 to 0.143], Standard Error of Mean 0.019 — Olo 10 mcg qd minus Placebo

15. Secondary Outcome: Trough FEV1 Response After 48 Weeks
Description: as for outcome 2
Time Frame: 1 h and 10 min prior to dose on the first day of randomized treatment (baseline) and -1 h (if available) and - 10 mins prior to study drug after 48 weeks
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 200 | 199 | 202
Liter | -0.74 (0.014) | 0.019 (0.014) | 0.017 (0.014)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.092, 95% CI [0.055 to 0.130], Standard Error of Mean 0.019 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.091, 95% CI [0.053 to 0.129], Standard Error of Mean 0.019 — Olo 10 mcg qd minus Placebo

16. Secondary Outcome: Peak FEV1 (0-3h) Response At Day 1
Description: Response was defined as change from baseline. Baseline peak FEV1 was defined as the mean of the available pre-dose peak FEV1 values prior to first dose of randomized treatment. Peak FEV1 (0-3h) values were obtained within 0 - 3 hours after treatment.
  Means are adjusted using a mixed effects model with treatment (trt), tio stratum, visit, trt-by- visit as fixed categorical effects, baseline and baseline-by-visit as fixed continuous covariates and patient as random effect.
Time Frame: as for outcome 4
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 208 | 206 | 206
Liter | 0.104 (0.015) | 0.259 (0.015) | 0.275 (0.015)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.155, 95% CI [0.115 to 0.194], Standard Error of Mean 0.020 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.171, 95% CI [0.131 to 0.211], Standard Error of Mean 0.020 — Olo 10 mcg qd minus Placebo

17. Secondary Outcome: Peak FEV1 (0-3h) Response After 2 Weeks
Description: Response was defined as change from baseline. Baseline peak FEV1 was defined as the mean of the available pre-dose peak FEV1 values prior to first dose of randomized treatment. Peak FEV1 (0-3h) values were obtained within 0 - 3 hours after treatment. Means are adjusted using a mixed effects model with treatment (trt), tio stratum, visit, trt-by-visit as fixed categorical effects, baseline and baseline-by-visit as fixed continuous covariates and patient as random effect.
Time Frame: as for outcome 5
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 208 | 206 | 206
Liter | 0.077 (0.015) | 0.254 (0.015) | 0.267 (0.015)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.177, 95% CI [0.137 to 0.217], Standard Error of Mean 0.020 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.190, 95% CI [0.150 to 0.230], Standard Error of Mean 0.020 — Olo 10 mcg qd minus Placebo

18. Secondary Outcome: Peak FEV1 (0-3h) Response After 6 Weeks
Description: as for outcome 17
Time Frame: 1 hour (h) and 10 minutes (min) prior to dose on the first day of randomized treatment (baseline) to -10 min, 5 min, 15 min, 30 min, 1 h, 2 h, and 3 h relative to dose after 6 weeks
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 208 | 206 | 206
Liter | 0.066 (0.015) | 0.238 (0.015) | 0.238 (0.015)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.172, 95% CI [0.132 to 0.212], Standard Error of Mean 0.021 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.172, 95% CI [0.132 to 0.212], Standard Error of Mean 0.021 — Olo 10 mcg qd minus Placebo

19. Secondary Outcome: Peak FEV1 (0-3h) Response After 12 Weeks
Description: as for outcome 17
Time Frame: 1 hour (h) and 10 minutes (min) prior to dose on the first day of randomized treatment (baseline) to -10 min, 5 min, 15 min, 30 min, 1 h, 2 h, and 3 h relative to dose after 12 weeks
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 208 | 206 | 206
Liter | 0.071 (0.015) | 0.235 (0.015) | 0.236 (0.015)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.164, 95% CI [0.123 to 0.204], Standard Error of Mean 0.021 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.165, 95% CI [0.124 to 0.206], Standard Error of Mean 0.021 — Olo 10 mcg qd minus Placebo

20. Secondary Outcome: Peak FEV1 (0-3h) Response After 24 Weeks
Description: as for outcome 17
Time Frame: as for outcome 7
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 208 | 206 | 206
Liter | 0.055 (0.016) | 0.230 (0.015) | 0.206 (0.015)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.175, 95% CI [0.134 to 0.216], Standard Error of Mean 0.021 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.151, 95% CI [0.110 to 0.192], Standard Error of Mean 0.021 — Olo 10 mcg qd minus Placebo

21. Secondary Outcome: Peak FEV1 (0-3h) Response After 48 Weeks
Description: as for outcome 17
Time Frame: as for outcome 8
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 208 | 206 | 206
Liter | 0.029 (0.016) | 0.198 (0.016) | 0.192 (0.016)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.169, 95% CI [0.128 to 0.211], Standard Error of Mean 0.021 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.163, 95% CI [0.121 to 0.205], Standard Error of Mean 0.021 — Olo 10 mcg qd minus Placebo

22. Secondary Outcome: Forced Vital Capacity (FVC) Area Under Curve 0-3 Hours (AUC 0-3h) Response At Day 1
Description: Response was defined as change from baseline. Baseline FVC was defined as the mean of the available pre-dose FVC values prior to the first dose of randomized treatment. Means are adjusted using a mixed effects model with treatment (trt), tio stratum, visit, trt-by-visit as fixed categorical effects, baseline and baseline-by-visit as fixed continuous covariates and patient as random effect. FVC AUC 0-3h was calculated using the trapezoidal rule, divided by the observation time to report in litres.
Time Frame: as for outcome 4
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 208 | 206 | 206
Liter | 0.063 (0.027) | 0.350 (0.027) | 0.392 (0.027)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.288, 95% CI [0.216 to 0.359], Standard Error of Mean 0.037 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.330, 95% CI [0.258 to 0.401], Standard Error of Mean 0.037 — Olo 10 mcg qd minus Placebo

23. Secondary Outcome: Forced Vital Capacity (FVC) Area Under Curve 0-3 Hours (AUC 0-3h) Response After 2 Weeks
Description: as for outcome 22
Time Frame: as for outcome 5
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 208 | 206 | 206
Liter | 0.026 (0.027) | 0.323 (0.027) | 0.353 (0.027)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.296, 95% CI [0.224 to 0.368], Standard Error of Mean 0.037 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.327, 95% CI [0.255 to 0.399], Standard Error of Mean 0.037 — Olo 10 mcg qd minus Placebo

24. Secondary Outcome: FVC Area Under Curve 0-3 Hours (AUC 0-3h) Response After 6 Weeks
Description: as for outcome 22
Time Frame: as for outcome 18
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 208 | 206 | 206
Liter | 0.022 (0.028) | 0.276 (0.028) | 0.316 (0.027)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.254, 95% CI [0.181 to 0.327], Standard Error of Mean 0.037 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.293, 95% CI [0.220 to 0.366], Standard Error of Mean 0.037 — Olo 10 mcg qd minus Placebo

25. Secondary Outcome: FVC Area Under Curve 0-3 Hours (AUC 0-3h) Response After 12 Weeks
Description: as for outcome 22
Time Frame: as for outcome 19
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 208 | 206 | 206
Liter | 0.003 (0.028) | 0.277 (0.028) | 0.295 (0.028)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.275, 95% CI [0.201 to 0.348], Standard Error of Mean 0.037 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.292, 95% CI [0.219 to 0.366], Standard Error of Mean 0.037 — Olo 10 mcg qd minus Placebo

26. Secondary Outcome: FVC Area Under Curve 0-3 Hours (AUC 0-3h) Response After 24 Weeks
Description: as for outcome 22
Time Frame: as for outcome 7
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 208 | 206 | 206
Liter | 0.026 (0.028) | 0.261 (0.028) | 0.281 (0.028)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.235, 95% CI [0.161 to 0.309], Standard Error of Mean 0.038 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.254, 95% CI [0.180 to 0.329], Standard Error of Mean 0.038 — Olo 10 mcg qd minus Placebo

27. Secondary Outcome: FVC Area Under Curve 0-3 Hours (AUC 0-3h) Response After 48 Weeks
Description: as for outcome 22
Time Frame: as for outcome 8
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 208 | 206 | 206
Liter | -0.040 (0.028) | 0.204 (0.028) | 0.231 (0.028)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.244, 95% CI [0.169 to 0.319], Standard Error of Mean 0.038 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.271, 95% CI [0.196 to 0.346], Standard Error of Mean 0.038 — Olo 10 mcg qd minus Placebo

28. Secondary Outcome: Trough FVC Response After 2 Weeks
Description: Response was defined as change from baseline. Baseline trough FVC was defined as the mean of the -1 hour and -10 minute measurements performed just prior to first dose of randomized treatment. Trough FVC is defined as the FVCs obtained at -10 mins prior to study drug inhalation as the end of the dosing interval or the mean of -1h and -10 min FVCs if both available. Means are adjusted using a mixed effects model with treatment (trt), tio stratum, visit, trt-by-visit as fixed categorical effects, baseline and baseline-by-visit as fixed continuous covariates and patient as random effect.
Time Frame: as for outcome 9
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 200 | 199 | 202
Liter | -0.015 (0.027) | 0.132 (0.027) | 0.169 (0.027)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.147, 95% CI [0.076 to 0.218], Standard Error of Mean 0.036 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.184, 95% CI [0.113 to 0.255], Standard Error of Mean 0.036 — Olo 10 mcg qd minus Placebo

29. Secondary Outcome: Trough FVC Response After 6 Weeks
Description: as for outcome 28
Time Frame: as for outcome 10
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 200 | 199 | 202
Liter | -0.005 (0.027) | 0.125 (0.027) | 0.135 (0.027)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0003, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.131, 95% CI [0.059 to 0.203], Standard Error of Mean 0.037 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.141, 95% CI [0.069 to 0.213], Standard Error of Mean 0.036 — Olo 10 mcg qd minus Placebo

30. Secondary Outcome: Trough FVC Response After 12 Weeks
Description: as for outcome 28
Time Frame: 1 h and 10 min prior to dose on the first day of randomized treatment (baseline) and -1 h (if available) and - 10 mins prior to study drug after 12 weeks
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 200 | 199 | 202
Liter | -0.030 (0.027) | 0.085 (0.027) | 0.130 (0.027)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0019, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.115, 95% CI [0.043 to 0.187], Standard Error of Mean 0.037 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.160, 95% CI [0.088 to 0.233], Standard Error of Mean 0.037 — Olo 10 mcg qd minus Placebo

31. Secondary Outcome: Trough FVC Response After 18 Weeks
Description: as for outcome 28
Time Frame: as for outcome 11
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 200 | 199 | 202
Liter | -0.028 (0.028) | 0.102 (0.027) | 0.134 (0.027)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0005, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.130, 95% CI [0.057 to 0.203], Standard Error of Mean 0.037 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.162, 95% CI [0.089 to 0.235], Standard Error of Mean 0.037 — Olo 10 mcg qd minus Placebo

32. Secondary Outcome: Trough FVC Response After 24 Weeks
Description: as for outcome 28
Time Frame: as for outcome 12
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 200 | 199 | 202
Liter | -0.028 (0.028) | 0.055 (0.027) | 0.096 (0.027)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0261, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.083, 95% CI [0.010 to 0.156], Standard Error of Mean 0.037 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0010, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.123, 95% CI [0.050 to 0.197], Standard Error of Mean 0.037 — Olo 10 mcg qd minus Placebo

33. Secondary Outcome: Trough FVC Response After 32 Weeks
Description: as for outcome 28
Time Frame: as for outcome 13
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 200 | 199 | 202
Liter | -0.026 (0.028) | 0.065 (0.028) | 0.097 (0.027)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0154, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.091, 95% CI [0.018 to 0.165], Standard Error of Mean 0.038 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0011, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.123, 95% CI [0.049 to 0.197], Standard Error of Mean 0.038 — Olo 10 mcg qd minus Placebo

34. Secondary Outcome: Trough FVC Response After 40 Weeks
Description: as for outcome 28
Time Frame: as for outcome 14
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 200 | 199 | 202
Liter | -0.044 (0.028) | 0.087 (0.028) | 0.111 (0.028)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0006, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.131, 95% CI [0.057 to 0.205], Standard Error of Mean 0.038 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.154, 95% CI [0.080 to 0.229], Standard Error of Mean 0.038 — Olo 10 mcg qd minus Placebo

35. Secondary Outcome: Trough FVC Response After 48 Weeks
Description: as for outcome 28
Time Frame: as for outcome 15
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 200 | 199 | 202
Liter | -0.083 (0.028) | 0.011 (0.028) | 0.032 (0.028)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0134, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.094, 95% CI [0.019 to 0.168], Standard Error of Mean 0.038 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0025, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.115, 95% CI [0.040 to 0.190], Standard Error of Mean 0.038 — Olo 10 mcg qd minus Placebo

36. Secondary Outcome: FVC Peak (0-3h) Response At Day 1
Description: Response was defined as change from baseline. Baseline FVC peak (0-3h) was defined as the mean of the available pre-dose FVC peak (0-3h) values prior to first dose of randomized treatment. FVC Peak (0-3h) values were obtained within 0 - 3 hours after treatment. Means are adjusted using a mixed effects model with treatment (trt), tio stratum, visit, trt-by-visit as fixed categorical effects, baseline and baseline-by-visit as fixed continuous covariates and patient as random effect.
Time Frame: as for outcome 4
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 208 | 206 | 206
Liter | 0.245 (0.029) | 0.509 (0.029) | 0.546 (0.029)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.263, 95% CI [0.187 to 0.339], Standard Error of Mean 0.039 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.300, 95% CI [0.225 to 0.376], Standard Error of Mean 0.039 — Olo 10 mcg qd minus Placebo

37. Secondary Outcome: FVC Peak (0-3h) Response After 2 Weeks
Description: as for outcome 36
Time Frame: as for outcome 5
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 208 | 206 | 206
Liter | 0.207 (0.029) | 0.471 (0.029) | 0.499 (0.029)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.264, 95% CI [0.188 to 0.341], Standard Error of Mean 0.039 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.292, 95% CI [0.216 to 0.368], Standard Error of Mean 0.039 — Olo 10 mcg qd minus Placebo

38. Secondary Outcome: FVC Peak (0-3h) Response After 6 Weeks
Description: as for outcome 36
Time Frame: as for outcome 18
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 208 | 206 | 206
Liter | 0.180 (0.029) | 0.430 (0.029) | 0.460 (0.029)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.251, 95% CI [0.174 to 0.328], Standard Error of Mean 0.039 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.280, 95% CI [0.203 to 0.358], Standard Error of Mean 0.039 — Olo 10 mcg qd minus Placebo

39. Secondary Outcome: FVC Peak (0-3h) Response After 12 Weeks
Description: as for outcome 36
Time Frame: as for outcome 19
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 208 | 206 | 206
Liter | 0.169 (0.029) | 0.421 (0.029) | 0.430 (0.029)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.251, 95% CI [0.174 to 0.329], Standard Error of Mean 0.040 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.260, 95% CI [0.183 to 0.338], Standard Error of Mean 0.040 — Olo 10 mcg qd minus Placebo

40. Secondary Outcome: FVC Peak (0-3h) Response After 24 Weeks
Description: as for outcome 36
Time Frame: as for outcome 7
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 208 | 206 | 206
Liter | 0.188 (0.030) | 0.419 (0.029) | 0.420 (0.030)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.232, 95% CI [0.153 to 0.310], Standard Error of Mean 0.040 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.232, 95% CI [0.154 to 0.311], Standard Error of Mean 0.040 — Olo 10 mcg qd minus Placebo

41. Secondary Outcome: FVC Peak (0-3h) Response After 48 Weeks
Description: as for outcome 36
Time Frame: as for outcome 8
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 208 | 206 | 206
Liter | 0.109 (0.030) | 0.356 (0.030) | 0.369 (0.030)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.247, 95% CI [0.168 to 0.327], Standard Error of Mean 0.040 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.260, 95% CI [0.181 to 0.340], Standard Error of Mean 0.041 — Olo 10 mcg qd minus Placebo

42. Secondary Outcome: Forced Vital Capacity (FVC) Area Under Curve 0-12 h (AUC 0-12h) Response at Day 85 (12 Weeks)
Description: Response was defined as change from baseline. Study baseline FVC was defined as the mean of the available pre-dose FVC values prior to the first dose of randomized treatment. Means are adjusted using a non-mixed effects model with treatment (trt), tio stratum, baseline as fixed effects. FVC AUC 0-12h was calculated from 0-12 hours post-dose using the trapezoidal rule, divided by the observation time (12h) to report in litres.
Time Frame: as for outcome 3
Population: Patients in FAS with spirometry data after 3 hours at Visit 5 (12-hour pulmonary function test set)
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 71 | 85 | 85
Liter | -0.019 (0.049) | 0.283 (0.045) | 0.230 (0.044)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, ANCOVA; Treatment, tiotropium stratum and baseline as fixed effects; Mean Difference (Final Values) = 0.302, 95% CI [0.181 to 0.422], Standard Error of Mean 0.061 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, ANCOVA; Treatment, tiotropium stratum and baseline as fixed effects; Mean Difference (Final Values) = 0.249, 95% CI [0.128 to 0.370], Standard Error of Mean 0.061 — Olo 10 mcg qd minus Placebo

43. Secondary Outcome: Weekly Mean Pre-dose Morning Peak Expiratory Flow Rate (PEF)
Description: Weekly mean pre-dose morning peak expiratory flow rate (PEF) at 48 weeks. PEFR measurements recorded by means of an e-Diary on a daily basis. This e-Diary was used to record the twice daily PEFs, study drug use, and rescue salbutamol (albuterol) use. The best of three readings for each measurement was recorded.
Time Frame: immediately upon arising (before drug administration) from Screening to week 48
Population: FAS
Measure: Mean (Standard Error); unit: L/min
Arm/Group | Placebo | Olodaterol (Olo) 5 mcg qd | Olodaterol (Olo) 10 mcg qd
Number analyzed (Participants) | 204 | 202 | 203
L/min | 180.019 (3.182) | 193.376 (3.207) | 195.475 (3.184)
Statistical Analysis 1: Comparison: Placebo vs Olodaterol (Olo) 5 mcg qd; Test type: Superiority or Other; p = 0.0018, ANCOVA; non-MMRM ANCOVA models by week, with treatment, tiotropium strata and baseline as fixed effects; Mean Difference (Final Values) = 13.357, 95% CI 2-sided [5.005 to 21.709], Standard Error of Mean 4.253
Statistical Analysis 2: Comparison: Placebo vs Olodaterol (Olo) 10 mcg qd; Test type: Superiority or Other; p = 0.0003, ANCOVA; non-MMRM ANCOVA models by week, with treatment, tiotropium strata and baseline as fixed effects; Mean Difference (Final Values) = 15.457, 95% CI 2-sided [7.114 to 23.800], Standard Error of Mean 4.248

44. Secondary Outcome: Weekly Mean Evening Peak Expiratory Flow Rate (PEF)
Description: Weekly mean evening peak expiratory flow rate (PEF) at 48 weeks. PEFR measurements recorded by means of an e-Diary on a daily basis. This e-Diary was used to record the twice daily PEFs, study drug use, and rescue salbutamol (albuterol) use. The best of three readings for each measurement was recorded.
Time Frame: at bedtime from Screening to week 48
Population: FAS
Measure: Mean (Standard Error); unit: L/min
Arm/Group | Placebo | Olodaterol (Olo) 5 mcg qd | Olodaterol (Olo) 10 mcg qd
Number analyzed (Participants) | 203 | 199 | 203
L/min | 190.676 (3.165) | 207.862 (3.202) | 205.236 (3.166)
Statistical Analysis 1: Comparison: Placebo vs Olodaterol (Olo) 5 mcg qd; Test type: Superiority or Other; p < 0.0001, ANCOVA; non-MMRM ANCOVA models by week, with treatment, tiotropium strata and baseline as fixed effects; Mean Difference (Final Values) = 17.186, 95% CI 2-sided [8.849 to 25.523], Standard Error of Mean 4.245
Statistical Analysis 2: Comparison: Placebo vs Olodaterol (Olo) 10 mcg qd; Test type: Superiority or Other; p = 0.0006, ANCOVA; non-MMRM ANCOVA models by week, with treatment, tiotropium strata and baseline as fixed effects; Mean Difference (Final Values) = 14.560, 95% CI 2-sided [6.259 to 22.860], Standard Error of Mean 4.226

45. Secondary Outcome: Weekly Mean Daytime Rescue Use
Description: The patient was to record in the e-Diary the number of puffs of salbutamol (albuterol) Metered-Dose Inhaler used each day and night.
Time Frame: From Screening to week 48
Population: FAS
Measure: Mean (Standard Error); unit: Number of puffs
Arm/Group | Placebo | Olodaterol (Olo) 5 mcg qd | Olodaterol (Olo) 10 mcg qd
Number analyzed (Participants) | 205 | 204 | 204
Number of puffs | 1.487 (0.136) | 0.967 (0.137) | 0.839 (0.136)
Statistical Analysis 1: Comparison: Placebo vs Olodaterol (Olo) 5 mcg qd; Test type: Superiority or Other; p = 0.0045, ANCOVA; non-MMRM ANCOVA models with treatment, tiotropium strata and baseline as fixed effects; Mean Difference (Final Values) = -0.520, 95% CI 2-sided [-0.878 to -0.162], Standard Error of Mean 0.182
Statistical Analysis 2: Comparison: Placebo vs Olodaterol (Olo) 10 mcg qd; Test type: Superiority or Other; p = 0.0004, ANCOVA; non-MMRM ANCOVA models with treatment, tiotropium strata and baseline as fixed effects; Mean Difference (Final Values) = -0.648, 95% CI 2-sided [-1.005 to -0.291], Standard Error of Mean 0.182

46. Secondary Outcome: Weekly Mean Nighttime Rescue Use
Description: as for outcome 45
Time Frame: From Screening to week 48
Population: FAS
Measure: Mean (Standard Error); unit: Number of puffs
Arm/Group | Placebo | Olodaterol (Olo) 5 mcg qd | Olodaterol (Olo) 10 mcg qd
Number analyzed (Participants) | 205 | 204 | 204
Number of puffs | 2.283 (0.151) | 1.701 (0.152) | 1.492 (0.152)
Statistical Analysis 1: Comparison: Placebo vs Olodaterol (Olo) 5 mcg qd; Test type: Superiority or Other; p = 0.0041, ANCOVA; non-MMRM ANCOVA models with treatment, tiotropium strata and baseline as fixed effects; Mean Difference (Final Values) = -0.582, 95% CI 2-sided [-0.979 to -0.185], Standard Error of Mean 0.202
Statistical Analysis 2: Comparison: Placebo vs Olodaterol (Olo) 10 mcg qd; Test type: Superiority or Other; p = 0.0001, ANCOVA; non-MMRM ANCOVA models with treatment, tiotropium strata and baseline as fixed effects; Mean Difference (Final Values) = -0.792, 95% CI 2-sided [-1.189 to -0.394], Standard Error of Mean 0.202

47. Secondary Outcome: Weekly Mean Daily (24h) Rescue Use
Description: as for outcome 45
Time Frame: From Screening to week 48
Population: FAS
Measure: Mean (Standard Error); unit: Number of puffs
Arm/Group | Placebo | Olodaterol (Olo) 5 mcg qd | Olodaterol (Olo) 10 mcg qd
Number analyzed (Participants) | 205 | 204 | 204
Number of puffs | 3.747 (0.265) | 2.642 (0.267) | 2.312 (0.265)
Statistical Analysis 1: Comparison: Placebo vs Olodaterol (Olo) 5 mcg qd; Test type: Superiority or Other; p = 0.0019, ANCOVA; non-MMRM ANCOVA models with treatment, tiotropium strata and baseline as fixed effects; Mean Difference (Final Values) = -1.104, 95% CI 2-sided [-1.799 to -0.409], Standard Error of Mean 0.354
Statistical Analysis 2: Comparison: Placebo vs Olodaterol (Olo) 10 mcg qd; Test type: Superiority or Other; p < 0.0001, ANCOVA; non-MMRM ANCOVA models with treatment, tiotropium strata and baseline as fixed effects; Mean Difference (Final Values) = -1.435, 95% CI 2-sided [-2.130 to -0.740], Standard Error of Mean 0.354

48. Secondary Outcome: Patient's Global Rating at Week 6
Description: Patients were asked to rate their respiratory condition relative to their condition prior to the first dose of study medication. The scale is a seven point scale: 1=very much better, 2=much better,3=a little better,4=no change,5=a little worse,6=much worse,7=very much worst.
Time Frame: Week 6 visit
Population: FAS
Measure: Mean (Standard Error); unit: Point on scale
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 189 | 194 | 197
Point on scale | 3.5 (0.1) | 3.0 (0.1) | 3.0 (0.1)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Model included treatment, tiotropium stratum, visit and treatment-by-visit interaction as fixed effects, patient as random; Mean Difference (Final Values) = -0.5, 95% CI [-0.7 to -0.3], Standard Error of Mean 0.1 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 48, analysis 1]; Mean Difference (Final Values) = -0.5, 95% CI [-0.7 to -0.3], Standard Error of Mean 0.1 — Olo 10 mcg qd minus Placebo

49. Secondary Outcome: Patient's Global Rating at Week 12
Description: as for outcome 48
Time Frame: Week 12 visit
Population: FAS
Measure: Mean (Standard Error); unit: Point on scale
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 189 | 194 | 197
Point on scale | 3.4 (0.1) | 3.0 (0.1) | 3.0 (0.1)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 48, analysis 1]; Mean Difference (Final Values) = -0.5, 95% CI [-0.7 to -0.2], Standard Error of Mean 0.1 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 48, analysis 1]; Mean Difference (Final Values) = -0.4, 95% CI [-0.6 to -0.2], Standard Error of Mean 0.1 — Olo 10 mcg qd minus Placebo

50. Secondary Outcome: Patient's Global Rating at Week 24
Description: as for outcome 48
Time Frame: Week 24 visit
Population: FAS
Measure: Mean (Standard Error); unit: Point on scale
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 189 | 194 | 197
Point on scale | 3.5 (0.1) | 3.0 (0.1) | 3.0 (0.1)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 48, analysis 1]; Mean Difference (Final Values) = -0.4, 95% CI [-0.7 to -0.2], Standard Error of Mean 0.1 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 48, analysis 1]; Mean Difference (Final Values) = -0.4, 95% CI [-0.7 to -0.2], Standard Error of Mean 0.1 — Olo 10 mcg qd minus Placebo

51. Secondary Outcome: Patient's Global Rating at Week 48
Description: as for outcome 48
Time Frame: Week 48 visit
Population: FAS
Measure: Mean (Standard Error); unit: Point on scale
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 189 | 194 | 197
Point on scale | 3.4 (0.1) | 3.1 (0.1) | 3.1 (0.1)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0109, Mixed Models Analysis; Model included treatment, tiotropium stratum,visit and treatment-by-visit interaction as fixed effects, patient as random; Mean Difference (Final Values) = -0.3, 95% CI [-0.5 to -0.1], Standard Error of Mean 0.1 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0031, Mixed Models Analysis; Model included treatment, tiotropium stratum visit and treatment-by-visit interaction as fixed effects, patient as random; Mean Difference (Final Values) = -0.3, 95% CI [-0.6 to -0.1], Standard Error of Mean 0.1 — Olo 10 mcg qd minus Placebo

52. Secondary Outcome: Time to First Chronic Obstructive Pulmonary Disease (COPD) Exacerbation
Description: Qualifying events of COPD were specifically pre-defined in the protocol. Other respiratory related events were evaluated by the investigator to see if they met the pre-defined criteria. Time to event was measured from the beginning of treatment. Cox regression analysis of treatment effect using tiotropium stratum as a stratification factor. Due to the limited number of events some statistics were not able to be calculated and are listed as N/A or are blank. The measure type is the First Quartile.
Time Frame: Baseline to end of study at 48 weeks.
Population: Treated set- all patients who received at least one dose of study medication
Measure: Mean (95% Confidence Interval); unit: days
Groups:
- Placebo (Tiotropium): Matching Placebo delivered by the Respimat Inhaler - tiotropium use stratum
- Placebo (Non-tiotropium): Matching Placebo delivered by the Respimat Inhaler - non-tiotropium use stratum.
- Olo 5 mcg qd (Tiotropium): Olodaterol 5 mcg qd (morning) delivered by the Respimat Inhaler - tiotropium stratum
- Olo 5 mcg qd (Non-tiotropium): Olodaterol 5 mcg qd (morning) delivered by the Respimat Inhaler - non-tiotropium stratum
- Olo 10 mcg qd (Tiotropium): Olodaterol 10 mcg qd (morning) delivered by the Respimat Inhaler - tiotropium stratum
- Olo 10 mcg qd(Non-tiotropium): Olodaterol 10 mcg qd (morning) delivered by the Respimat Inhaler - non-tiotropium stratum
Arm/Group | Placebo (Tiotropium) | Placebo (Non-tiotropium) | Olo 5 mcg qd (Tiotropium) | Olo 5 mcg qd (Non-tiotropium) | Olo 10 mcg qd (Tiotropium) | Olo 10 mcg qd(Non-tiotropium)
Number analyzed (Participants) | 49 | 160 | 47 | 161 | 51 | 156
days | 194.0 [29.0 to 305.0] | 160.0 [139.0 to 204.0] | 203.0 [76.0 to NA] — N/A indicates this statistic was not available due to the low number of events observed. | 236.0 [158.0 to 337.0] | 167.0 [74.0 to NA] — N/A indicates this statistic was not available due to the low number of events observed. | 239.0 [192.0 to 306.0]
Statistical Analysis 1: Comparison: Placebo (Tiotropium) vs Placebo (Non-tiotropium) vs Olo 5 mcg qd (Tiotropium) vs Olo 5 mcg qd (Non-tiotropium); Test type: Superiority or Other; p = 0.0658, Regression, Cox; Model included a stratification factor for tiotropium use stratum and a covariate for treatment group; Hazard Ratio (HR) = 0.728, 95% CI 2-sided [0.522 to 1.016], Standard Error of Mean 0.124 — Comparison of Olo 5 mcg qd to placebo across stratum
Statistical Analysis 2: Comparison: Placebo (Tiotropium) vs Placebo (Non-tiotropium) vs Olo 10 mcg qd (Tiotropium) vs Olo 10 mcg qd(Non-tiotropium); Test type: Superiority or Other; p = 0.1701, Regression, Cox; Model included a stratification factor for tiotropium use stratum and a covariate for treatment group; Hazard Ratio (HR) = 0.799, 95% CI 2-sided [0.576 to 1.107], Standard Error of Mean 0.133 — Comparison of Olo 10 mcg qd to placebo across stratum

53. Secondary Outcome: Time to First Chronic Obstructive Pulmonary Disease (COPD) Exacerbation Leading to Hospitalization
Description: Qualifying events of COPD were specifically pre-defined in the protocol. Other respiratory related events were evaluated by the investigator to see if they met the pre-defined criteria. These exacerbations required hospitalization. Time to event was measured from the beginning of treatment. Cox regression analysis of treatment effect using tiotropium stratum as a stratification factor. Due to the limited number of events some statistics were not able to be calculated and are listed as N/A or are blank. The measure type is the First Quartile.
Time Frame: Baseline to end of study at 48 weeks.
Population: Treated set- all patients who received at least one dose of study medication
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Placebo (Tiotropium) | Placebo (Non-tiotropium) | Olo 5 mcg qd (Tiotropium) | Olo 5 mcg qd (Non-tiotropium) | Olo 10 mcg qd (Tiotropium) | Olo 10 mcg qd(Non-tiotropium)
Number analyzed (Participants) | 49 | 160 | 47 | 161 | 51 | 156
days | NA [NA to NA] — N/A indicates this statistic was not available due to the low number of events observed. | NA [NA to NA] — N/A indicates this statistic was not available due to the low number of events observed. | NA [NA to NA] — N/A indicates this statistic was not available due to the low number of events observed. | NA [NA to NA] — N/A indicates this statistic was not available due to the low number of events observed. | NA [NA to NA] — N/A indicates this statistic was not available due to the low number of events observed. | NA [344.0 to NA] — N/A indicates this statistic was not available due to the low number of events observed.
Statistical Analysis 1: Comparison: Placebo (Tiotropium) vs Placebo (Non-tiotropium) vs Olo 5 mcg qd (Tiotropium) vs Olo 5 mcg qd (Non-tiotropium); Test type: Superiority or Other; p = 0.2754, Regression, Cox; Model included a stratification factor for tiotropium use stratum and a covariate for treatment group; Hazard Ratio (HR) = 0.656, 95% CI 2-sided [0.313 to 1.374], Standard Error of Mean 0.247 — Comparison of Olo 5 mcg qd to placebo across stratum
Statistical Analysis 2: Comparison: Placebo (Tiotropium) vs Placebo (Non-tiotropium) vs Olo 10 mcg qd (Tiotropium) vs Olo 10 mcg qd(Non-tiotropium); Test type: Superiority or Other; p = 0.9792, Regression, Cox; Model included a stratification factor for tiotropium use stratum and a covariate for treatment group; Hazard Ratio (HR) = 1.010, 95% CI 2-sided [0.521 to 1.961], Standard Error of Mean 0.342 — Comparison of Olo 10 mcg qd to placebo across stratum

54. Secondary Outcome: Time to First Moderate Chronic Obstructive Pulmonary Disease (COPD) Exacerbation
Description: Qualifying events of COPD were specifically pre-defined in the protocol. Other respiratory related events were evaluated by the investigator to see if they met the pre-defined criteria. These exacerbations did not lead to hospitalization but included treatment with antibiotics and/or systemic steroids. Time to event was measured from the beginning of treatment. Cox regression analysis of treatment effect using tiotropium stratum as a stratification factor. Due to the limited number of events some statistics were not able to be calculated and are listed as N/A or are blank. The measure type is the First Quartile.
Time Frame: Baseline to end of study at 48 weeks.
Population: Treated set- all patients who received at least one dose of study medication
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Placebo (Tiotropium) | Placebo (Non-tiotropium) | Olo 5 mcg qd (Tiotropium) | Olo 5 mcg qd (Non-tiotropium) | Olo 10 mcg qd (Tiotropium) | Olo 10 mcg qd(Non-tiotropium)
Number analyzed (Participants) | 49 | 160 | 47 | 161 | 51 | 156
days | 194.0 [29.0 to 305.0] | 216.0 [158.0 to NA] — N/A indicates this statistic was not available due to the low number of events observed. | 218.0 [76.0 to NA] — N/A indicates this statistic was not available due to the low number of events observed. | 344.0 [206.0 to NA] — N/A indicates this statistic was not available due to the low number of events observed. | 170.0 [74.0 to NA] — N/A indicates this statistic was not available due to the low number of events observed. | 309.0 [220.0 to NA] — N/A indicates this statistic was not available due to the low number of events observed.
Statistical Analysis 1: Comparison: Placebo (Tiotropium) vs Placebo (Non-tiotropium) vs Olo 5 mcg qd (Tiotropium) vs Olo 5 mcg qd (Non-tiotropium); Test type: Superiority or Other; p = 0.1194, Regression, Cox; Model included a stratification factor for tiotropium use stratum and a covariate for treatment group; Hazard Ratio (HR) = 0.739, 95% CI 2-sided [0.506 to 1.078], Standard Error of Mean 0.142 — Comparison of Olo 5 mcg qd to placebo across stratum
Statistical Analysis 2: Comparison: Placebo (Tiotropium) vs Placebo (Non-tiotropium) vs Olo 10 mcg qd (Tiotropium) vs Olo 10 mcg qd(Non-tiotropium); Test type: Superiority or Other; p = 0.2570, Regression, Cox; Model included a stratification factor for tiotropium use stratum and a covariate for treatment group; Hazard Ratio (HR) = 0.811, 95% CI 2-sided [0.561 to 1.174], Standard Error of Mean 0.153 — Comparison of Olo 10 mcg qd to placebo across stratum

55. Secondary Outcome: Number of COPD Exacerbations
Description: Qualifying events of COPD were specifically pre-defined in the protocol. Other respiratory related events were evaluated by the investigator to see if they met the pre-defined criteria.
Time Frame: Baseline to end of study at week 48 visit
Population: Treated set- all patients who received at least one dose of study medication
Measure: Mean (Standard Error); unit: Number of COPD exacerbations
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 209 | 208 | 207
Number of COPD exacerbations | 0.7476 (0.0972) | 0.5842 (0.0791) | 0.6322 (0.0822)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.1631, Negative binomial regression; Regression of treatment effect using tiotropium strata as a covariate, a log link function and log(exposure) as offset; Incidence rate ratio = 0.7815, 95% CI 2-sided [0.5524 to 1.1054], Standard Error of Mean 0.1380 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.3342, Negative binomial regression; Regression of treatment effect using tiotropium strata as a covariate, a log link function and log(exposure) as offset; Incidence rate ratio = 0.8456, 95% CI 2-sided [0.6015 to 1.1889], Standard Error of Mean 0.1467 — Olo 10 mcg qd minus Placebo

56. Secondary Outcome: Number of COPD Exacerbations Requiring Hospitalization
Description: Qualifying events of COPD were specifically pre-defined in the protocol. Other respiratory related events were evaluated by the investigator to see if they met the pre-defined criteria. These exacerbations required hospitalization.
Time Frame: Baseline to end of study at week 48 visit
Population: Treated set- all patients who received at least one dose of study medication
Measure: Mean (Standard Error); unit: Number of COPD exacerbations
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 209 | 208 | 207
Number of COPD exacerbations | 0.1010 (0.0314) | 0.0662 (0.0224) | 0.1133 (0.0319)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.2985, Negative binomial regression; Regression of treatment effect using tiotropium strata as a covariate, a log link function and log(exposure) as offset; Incidence rate ratio = 0.6550, 95% CI 2-sided [0.2947 to 1.4556], Standard Error of Mean 0.2664 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.7550, Negative binomial regression; Regression of treatment effect using tiotropium strata as a covariate, a log link function and log(exposure) as offset; Incidence rate ratio = 1.1211, 95% CI 2-sided [0.5464 to 2.3003], Standard Error of Mean 0.4103 — Olo 10 mcg qd minus Placebo

57. Secondary Outcome: Number of Moderate Chronic Obstructive Pulmonary Disease (COPD) Exacerbations
Description: Qualifying events of COPD were specifically pre-defined in the protocol. Other respiratory related events were evaluated by the investigator to see if they met the pre-defined criteria. These exacerbations did not lead to hospitalization but included treatment with antibiotics and/or systemic steroids.
Time Frame: Baseline to end of study at 48 weeks.
Measure: Mean (Standard Error); unit: Number of COPD exacerbations
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 209 | 208 | 207
Number of COPD exacerbations | 0.5745 (0.0844) | 0.4643 (0.0714) | 0.4875 (0.0723)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.2911, Negative binomial regression; Regression of treatment effect using tiotropium strata as a covariate, a log link function and log(exposure) as offset; Incidence rate ratio = 0.8081, 95% CI 2-sided [0.5438 to 1.2008], Standard Error of Mean 0.1630 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.4086, Negative binomial regression; Regression of treatment effect using tiotropium strata as a covariate, a log link function and log(exposure) as offset; Incidence rate ratio = 0.8485, 95% CI 2-sided [0.5743 to 1.2535], Standard Error of Mean 0.1686 — Olo 10 mcg qd minus Placebo

58. Secondary Outcome: Changes in Safety Parameters Related to Treatment
Description: Occurrence of bronchoconstriction, cardiac disorders and investigations related to treatment. Bronchoconstriction is defined as any of the following events: Drop in trough FEV1 >= 15%, Rescue medication use within 30 min of inhaling randomized treatment on a clinic test day or Cough, wheeze, or dyspnoea AE within 30 min of inhaling randomized treatment on a clinic test day.
Time Frame: 48 weeks
Population: Treated set.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 209 | 208 | 207
percentage of participants
  Bronchoconstriction | 13.4 | 2.4 | 3.9
  Atrial fibrillation | 0.0 | 0.0 | 1.0
  Angina pectoris | 0.0 | 0.5 | 0.0
  Ventricular extrasystoles | 0.0 | 0.5 | 0.0
  Electrocardiogram QT prolonged | 0.5 | 0.5 | 0.0
  Forced expiratory volume decreased | 0.0 | 0.0 | 0.5

59. Secondary Outcome: Change From Baseline in Potassium
Description: Laboratory testing: Average change from baseline of potassium measured. The laboratory tests at Day 1 were considered the baseline measurements.
Time Frame: Day 1 and at 12, 24 and 48 weeks
Population: Treated set.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | Olodaterol (Olo) 5 mcg qd | Olodaterol (Olo) 10 mcg qd
Number analyzed (Participants) | 197 | 201 | 201
mmol/L | 0.0 (0.4) | 0.0 (0.3) | 0.0 (0.3)

ADVERSE EVENTS:
Time Frame: 48 weeks
Groups:
- Olo 5 mcg: Olodaterol 5 mcg qd (morning) delivered by the Respimat Inhaler.
- Olo 10 mcg: Olodaterol 10 mcg qd (morning) delivered by the Respimat Inhaler.
Arm/Group | Placebo | Olo 5 mcg | Olo 10 mcg
Serious Adverse Events (participants affected / at risk) | 34/209 | 39/208 | 43/207
Other Adverse Events (participants affected / at risk) | 93/209 | 83/208 | 78/207
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=209) | Olo 5 mcg (N=208) | Olo 10 mcg (N=207)
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 0
Angina unstable (Cardiac disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 2
Atrioventricular block complete (Cardiac disorders) | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 0 | 0
Cor pulmonale acute (Cardiac disorders) | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1 | 1
Coronary artery occlusion (Cardiac disorders) | 2 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Right ventricular failure (Cardiac disorders) | 0 | 0 | 1
Goitre (Endocrine disorders) | 0 | 0 | 1
Amaurosis fugax (Eye disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Colonic polyp (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 2 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatic mass (Gastrointestinal disorders) | 0 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 1
Bone abscess (Infections and infestations) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 1 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 | 1 | 0
Lobar pneumonia (Infections and infestations) | 1 | 1 | 1
Lung infection (Infections and infestations) | 0 | 1 | 0
Orchitis (Infections and infestations) | 1 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 1 | 1
Pneumonia (Infections and infestations) | 4 | 2 | 2
Pulmonary tuberculosis (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 2 | 0
Arterial restenosis (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 2
Fracture displacement (Injury, poisoning and procedural complications) | 1 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 0
Neck injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 | 0 | 1
Skeletal injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1
Myoglobin blood increased (Investigations) | 0 | 0 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Spinal cord neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Basal ganglia haemorrhage (Nervous system disorders) | 0 | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 2
Cervical myelopathy (Nervous system disorders) | 0 | 1 | 0
Epidural lipomatosis (Nervous system disorders) | 0 | 0 | 1
Hemiplegia (Nervous system disorders) | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 2
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0
Bipolar disorder (Psychiatric disorders) | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 14 | 10 | 18
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Aortic aneurysm (Vascular disorders) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0
Femoral arterial stenosis (Vascular disorders) | 0 | 1 | 0
Hypertensive crisis (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=209) | Olo 5 mcg (N=208) | Olo 10 mcg (N=207)
Bronchitis (Infections and infestations) | 8 | 11 | 6
Nasopharyngitis (Infections and infestations) | 13 | 21 | 13
Upper respiratory tract infection (Infections and infestations) | 15 | 21 | 13
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 57 | 40 | 49
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 14 | 7
Hypertension (Vascular disorders) | 12 | 3 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication